CLINICAL TRIAL: NCT04645940
Title: A Phase 1, Open-Label, 3 Period, Randomized 2-Sequence Study to Evaluate the Effect of Food and Rabeprazole, a Proton Pump Inhibitor, on the Pharmacokinetics of Fruquintinib in Healthy Subjects
Brief Title: Fruquintinib Food Effect and Proton Pump Inhibitor Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-013-00US1
Record Dates: First submitted 2020-10-26; First posted 2020-11-27 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2020-10

CONDITIONS: Drug Interaction; Food-drug Interaction
MeSH Terms: interventions — HMPL-013; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fed/Fasted (Experimental): fruquintinib 5 mg with food on Day 1 and fruquintinib 5 mg without food on Day 15. 40 mg rabeprazole from Day 23 to Day 29. On Day 29, fruquintinib 5 mg one hour after rabeprazole dose.
  Interventions: Drug: fruquintinib with food/fruquintinib without food/fruquintinib with rabeprazole
- Fasted/Fed (Experimental): fruquintinib 5 mg without food on Day 1 and fruquintinib 5 mg with food on Day 15. 40 mg rabeprazole from Day 23 to Day 29. On Day 29, fruquintinib 5 mg one hour after rabeprazole dose.
  Interventions: Drug: fruquintinib without food/fruquintinib with food/fruquintinib with rabeprazole

INTERVENTIONS:
Drug: fruquintinib with food/fruquintinib without food/fruquintinib with rabeprazole — fruquintinib 5 mg with food on Day 1 and fruquintinib 5 mg without food on Day 15.
  40 mg rabeprazole from Day 23 to Day 28. 40 mg rabeprazole one hour before 5 mg fruquintinib Day 29.
  Other Names: HMPL-013; rabeprazole 40 mg
  Arms: Fed/Fasted
Drug: fruquintinib without food/fruquintinib with food/fruquintinib with rabeprazole — fruquintinib 5 mg without food on Day 1 and fruquintinib 5 mg with food on Day 15.
  40 mg rabeprazole from Day 23 to Day 28. 40 mg rabeprazole one hour before 5 mg fruquintinib Day 29.
  Other Names: HMPL-013; rabeprazole 40 mg
  Arms: Fasted/Fed

SUMMARY:
The purpose of this is to evaluate the effect of food and the effect of a proton pump inhibitor (rabeprazole) on the pharmacokinetics of fruquintinib.

DETAILED DESCRIPTION:
This study will be a single center, open label, 3-period, randomized 2-sequence study conducted with 14 healthy male or female subjects. The study will consist of a Screening Phase (Screening and Day -1), a Treatment Phase (Periods 1, 2, and 3), and an End of Study (EOS) Phase. For Periods 1 and 2, subjects will be randomized into 1 of the 2 treatment sequences, with all subjects then moving to the same treatment in Period 3.

Periods 1 and 2: 14 subjects will be randomly assigned in a 1:1 ratio to 1 of 2 possible treatment sequences:

* Fed/Fasted: fruquintinib 5 mg with food on Day 1 and fruquintinib 5 mg without food on Day 15
* Fasting/Fed: fruquintinib 5 mg without food on Day 1 and fruquintinib 5 mg with food on Day 15

Period 3: all subjects will take rabeprazole 40 mg orally once daily in the morning from Day 23 to Day 29. On the morning of Day 29, all subjects will take rabeprazole 40 mg orally without food one hour before taking a fruquintinib 5 mg oral dose. Subjects will continue to fast until lunch.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking, healthy male or female between the ages of 18 and 55 years (inclusive) at the time of informed consent.
2. Body mass index (BMI) > 18 and ≤ 29 kg/m2 at Screening.
3. Females must be of non-childbearing potential (eg, postmenopausal [defined as cessation of all menstrual periods for at least 1 year confirmed by follicle-stimulating hormone (FSH) test ≥ 40 UI/L] or surgically sterile by total hysterectomy, bilateral oophorectomy, or bilateral tubal ligation).
4. Males who have not had a successful vasectomy and are partners of women of childbearing potential must use, or their partners must use, a medically acceptable method of contraception starting for at least 1 menstrual cycle prior to and throughout the entire study period, and for 2 weeks after the last dose of study drug. Those with partners using hormonal contraceptives must also use an additional approved method of contraception, such as a condom with spermicide. Males who have had a successful vasectomy (confirmed azoospermia, documentation needed) require no additional contraception. No sperm donation is allowed during the study period and for 90 days after study drug discontinuation.

Exclusion Criteria:

1. Evidence of clinically significant cardiovascular, hepatic, gastrointestinal (GI), renal, respiratory, endocrine, hematological, neurological, or psychiatric disease or abnormalities.
2. History of any GI surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, history of stomach or intestinal surgery or resection, except appendectomy and hernia repair will be allowed).
3. Clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
4. Food allergy deemed clinically significant per PI.
5. Clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at Screening or Day -1 Check-in (baseline).
6. Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at Screening or Day -1 Check-in (baseline).
7. Clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval > 480 msec), or has a family history of prolonged QTc syndrome or sudden death.
8. Gilbert's syndrome as indicated by total bilirubin >upper limit of normal (ULN) and subsequent measurement of direct bilirubin is not within normal range.
9. History of smoking or use of nicotine-containing substances within the previous 2 months, as determined by medical history or subject's verbal report and confirmed by cotinine test at Screening and Check-In for any one of the treatment periods.
10. History of drug or alcohol misuse within 6 months prior to Screening or a positive urine drug test at Screening or Check-in for any one of the treatment periods.
11. Diagnosed with acquired immune deficiency syndrome (AIDS) or has performed tests that are positive for human immunodeficiency virus (HIV), Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
12. Participated in a clinical study of other drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the subject is currently enrolled in another clinical study.
13. Consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
14. Consumed herbal preparations/medications, including, but not limited to kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose.
15. Weight loss or gain of > 10% within 4 weeks prior to the first dose.
16. Received blood or blood products within 4 weeks, or donated blood or blood products within 8 weeks prior to the first dose or donated double red cell within 16 weeks prior to first dose.
17. Used any over-the-counter (OTC) medications or prescription drugs within 2 weeks prior to the first dose.
18. Used CYP3A inducers (including St. John's wort) or inhibitors within 2 weeks before Day 1.
19. Allergic to any of the study drugs or to any of their excipients.
20. Used a PPI within 4 days prior to the first dose or a histamine 2 (H2) receptor antagonist (H2 blocker) within 2 days prior to the first dose.
21. Cannot abstain from using a PPI or an H2 blocker or locally acting antacids (eg, Gaviscon, Gelusil, Maalox, Milk of Magnesia, Mylanta, Rolaids, Tums).
22. Any condition that would make him or her, in the opinion of the investigator or sponsor, unsuitable for the study, or who, in the opinion of the investigator, is not likely to complete the study for any reason.
23. Female subject is pregnant, lactating, or breastfeeding.
24. Cannot consume study designed high-fat meal due to diet restrictions or being vegetarian/vegan.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
AUC(0-t) of fruquintinib: area under the plasma-concentration time curve from time 0 to time of the last measurable concentration | Up to 36 days
  Pharmacokinetics of fruquintinib by assessment of area under the plasma concentration time curve from zero to the last measurable concentration
AUC(0-inf) of fruquintinib | up to 36 days
  Pharmacokinetics of fruquintinib by assessment of area under the plasma concentration curve from zero extrapolated to infinity (if data permit)
Cmax of fruquintinib | up to 36 days
  Pharmacokinetics of fruquintinib by assessment of maximum plasma fruquintinib concentration

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events as assessed by CTCAE v5.0 | up to 36 days
  To evaluate the safety, in healthy subjects, of a single dose of 5 mg fruquintinib administered fed or fasted and with rabeprazole

CONTACTS AND LOCATIONS:
Overall Officials: Youngiun Kim, MD, Principal Investigator — WCCT Global Inc
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No